CLINICAL TRIAL: NCT01259531
Title: A 12-week, Open Label, Multi-center Study to Investigate the Efficacy and Safety of a α1A Adrenoceptor Selective Antagonist Silodosin on Urinary Disturbance Associated With Benign Prostatic Hyperplasia
Brief Title: Study of a α1A Adrenoceptor Selective Antagonist Silodosin to Treat Severe Benign Prostatic Hyperplasia(BPH)
Acronym: STRONG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Collaborators: Chonnam National University Hospital (Other); Kangdong Sacred Heart Hospital (Other); Yeungnam University Hospital (Other); Pusan National University Hospital (Other); Seoul National University Hospital (Other); Samsung Medical Center (Other); Seoul St. Mary's Hospital (Other); Korea University Guro Hospital (Other); Chonbuk National University Hospital (Other); Asan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWP-SDS-403
Record Dates: First submitted 2010-12-07; First posted 2010-12-14 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: strong; silodosin; benign prostatic hyperplasia; BPH; lower urinary tract symptoms associated with severe BPH
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — silodosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Silodosin (Experimental): Silodosin will be administered during 12 weeks, 8 mg (4 mg x 2 cap) QD with morning meal.
  Interventions: Drug: Silodosin

INTERVENTIONS:
Drug: Silodosin — Silodosin will be administered during 12 weeks, 8 mg (4 mg x 2 cap) QD with morning meal.
  Other Names: Brand name in Korea : THRUPAS

SUMMARY:
This clinical study is designed to evaluate the efficacy and safety of silodosin in a 12 week treatment of patients with severe urinary disorders associated with benign prostatic hyperplasia (BPH).

ELIGIBILITY:
Inclusion Criteria:

* Is at least 50 years old
* Has a urinary disturbance associated with severe BPH and has a total IPSS score 20 or higher
* Has a QoL score of 3 or higher
* Has a urine volume of 120mL or greater and a Qmax of below 15mL/sec
* Has a PRV of below 100mL
* Voluntarily decides to participate in this trial and sign with informed consent form

Exclusion Criteria:

* Has been administered silodosin
* Has been administered an α1A-adrenoceptor blocker within one month
* Has been prescribed antiandrogens except 5α-reductase inhibitors within a year
* Has had phytotherapy within 3 months
* Has had prostatectomy
* Has had intrapelvic radiation therapy
* Has had transurethral microwave hyperthermia of transurethral needle ablation
* Is suspected to have implications that are likely to affect urine passing such as neurogenic bladder, bladder calculus or active urinary tract infection (UTI).
* Is conducting self-catherterization
* Has a renal impairment with a serum creatinine of 2.0mg/dL or greater
* Has severe hepatic disorders (hepatic insufficiency, cirrhosis, jaundice, hepatoma) or has a total bilirubin of 2.5mg/dl or higher or has AST/ALT 2.5 times higher than the normal (upper) level
* Has suffered from a severe arrhythmia, cardiac failure, cardiac infarction, unstable angina, cerebral infarction within 6 months
* Has experienced allergy to α1 receptor blockers
* Has orthostatic hypotension around the time of Screening Visit
* Has participated in other clinical trials within 8 weeks prior to Screening Visit
* Has a Prostate specific antigen(PSA) of higher 10ng/mL or has been diagnosed with tumor identified by a biopsy even though he has a PSA of lower 10ng/mL (Patient who has been administered 5α-reductase inhibitors for more than 3 months are presumed to have 2 times higher than their actual PSA levels)
* Has been taking unstable dosing of 5α-reductase inhibitors like finasteride or dutasteride for the past 3 months or is expected to change the dosage during the trial.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Total International prostate symptom score(IPSS) score before and after treatment | For 12 weeks
  Assess the improvement of lower urinary tract symptoms with change in total IPSS score before and after treatment.

SECONDARY OUTCOMES:
Quality of life(QoL) score before and after treatment | For 12 weeks
  Assess the improvement of lower urinary tract symptoms with change in QoL score before and after treatment.
Maximal urinary flow rate(Qmax) before and after treatment | For 12 weeks
  Assess the improvement of lower urinary tract symptoms with change in Qmax before and after treatment.
Voiding score of IPSS before and after treatment | For 12 weeks
  Assess the improvement of lower urinary tract symptoms with change in voiding scores before and after treatment.
Storage scores of IPSS before and after treatment | For 12 weeks
  Assess the improvement of lower urinary tract symptoms with change in storage scores before and after treatment.
Post void residual urine volume(PVR) before and after treatment | For 12 weeks
  Assess the improvement of lower urinary tract symptoms with change in post void residual urine volume(PRV) before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: G.S. Park, Prof, Study Chair — Chonnam National Univ.; D.Y. Yang, Prof, Principal Investigator — Kangdong Sacred Heart; K.H. Moon, Prof, Principal Investigator — Yeongnam Univ. Medical; N.C. Park, Principal Investigator — Pusan National Univ. Hospital; S.W. Kim, Prof, Principal Investigator — Seoul National Univ. Hospital; S.W. Lee, Prof, Principal Investigator — Samsung Medical Center; S.W. Kim, Prof, Principal Investigator — Seoul St. Mary's Hospital; D.G. Moon, Prof, Principal Investigator — Korea Univ. Guro Hospital; J.K. Park, Prof, Principal Investigator — Chunbuk National Univ. Hospital; T.Y. Ahn, Prof, Principal Investigator — Asan Medical Center
Locations (1):
- Seoul national university hospital, Seoul, South Korea